CLINICAL TRIAL: NCT01381796
Title: A Phase I, Single Center, Open Label, Randomized, Single-Dose, Three-Way Crossover Study to Compare the Pharmacokinetics and Bioavailability of Two NP101 (Sumatriptan Iontophoretic Transdermal Patch) With an Oral Formulation of Imitrex in Healthy Volunteers and to Collect Resistance Data During Application of NP101
Brief Title: Compare PK and Bioavailability of 2 NP101 Patches With Oral Imitrex in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PROT-15-NP101-013
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Compare Bioequivalence Patches Previously Used in the NP101-007 Study
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A - NP101 (Active Comparator)
  Interventions: Drug: NP101
- Treatment C - oral sumatriptan succinate (Active Comparator)
  Interventions: Drug: sumatriptan succinate
- Treatment B - NP101B (Experimental)
  Interventions: Drug: NP101
- Treatment D - NP101D (Experimental)
  Interventions: Drug: NP101

INTERVENTIONS:
Drug: NP101 — comparison of NP101 with minor patch modifications
  Arms: Treatment A - NP101; Treatment B - NP101B; Treatment D - NP101D
Drug: sumatriptan succinate — tablet, 100 mg
  Other Names: Imitrex
  Arms: Treatment C - oral sumatriptan succinate

SUMMARY:
The purpose of this research is to:

1. Compare two study patches having minor differences in patch components
2. Compare the pharmacokinetics (PK - how the body absorbs, metabolizes and eliminates medication) of NP101 (study patches) versus a currently approved oral formulation of Imitrex
3. Collect resistance data during application of NP101 (study patch)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects, between the ages of 18 to 65 years, at the time of screening.
* Subject judged to be in good health, base upon result of medical history, physical examination, vital signs, ECG and laboratory profile. Subjects will not have any clinically significant abnormal laboratory parameters, vital signs or ECG parameters in order to qualify for enrollment.
* Subject must be capable of reading and understanding English or Spanish, and be able to carry-out all study procedures, and voluntarily sign and date an informed consent (IC) agreement approved by an IRB.
* Subject must have a negative drug screen.
* Subject has two acceptable patch application sites (left and/or right upper arms) that is relatively hair free and has no scars, tattoos, scratches or bruises.
* Subjects must have body mass index of 18 to 25 kg/m2 inclusive.
* Subjects must be nonsmokers, defined as having not used any tobacco products in the 6 months before screening.
* Subjects must have not consumed alcoholic beverages, poppy seeds, grapefruit, and/or grapefruit juice within 72 hours prior to admission to the clinic for Period 1 and for the duration of the study.
* Subjects must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.
* The subject must be likely to complete the entire study.

Exclusion Criteria:

* Subject has suspected or confirmed cardiovascular disease that contraindicates study participation.
* Subject has a history of epilepsy or conditions associated with a lowered seizure threshold.
* Subject with Raynaud's disease.
* Subject has a history of basilar or hemiplegic migraines.
* Subject has a current diagnosis of a major depressive disorder per the Diagnostic and Statistical Manual of Mental Disorders version 4 revised (DSM-IV-R).
* Subject has taken non-triptan serotonergic drugs including selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs, including Wellbutrin), tricyclic antidepressants (TCAs), monoamine oxidase inhibitors (MAOIs) or preparations containing St. Joh's Wort within 1 month prior to screening and/or is planning to start any of these medications during the study and through the End of Study visit.
* Subject is unwilling to discontinue use of a phosphodiesterase type 5 inhibitor (e.g. Viagra, Levitra, or Cialis) from screening through the End of Study visit.
* Subject with a history of a significant allergy or hypersensitivity to any component of the study patch used in this study (NP101 formulation details can be found in the NP101 Investigator Brochure).
* Subject who has any generalized skin irritation or disease including eczema, psoriasis, melanoma, acne or contact dermatitis.
* Subject is positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Subject has hepatic dysfunction defined as SGOT/AST or SGPT/ALT greater than or equal to 2 times the upper limit of normal (ULN)range, or alkaline phosphatase or total bilirubin greater than or equal to 1.5 times the ULN range or if in the opinion of the Investigator the subject's history, physical examination or other laboratory tests suggest hepatic dysfunction.
* Female subjects who are pregnant, breast feeding, or if of childbearing potential, is not using or is unwilling to use an effective form of contraception during the study and for a period of 30 days following final dosing. Acceptable methods of contraception include barrier method with spermicide, intrauterine device (IUD), steroidal contraceptive (oral, transdermal, implanted or injected) or abstinence. If the exclusive male partner is surgically sterile, this will be acceptable.
* Subject has known history of tolerability issues with sumatriptan.
* Subject who is considered by investigator or NuPathe, for any reason, to be an unsuitable candidate for this study.
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence.
* Subject has participated in a clinical study within 30 days of screening.
* Subject has clinically significant abnormal laboratory parameters, vial signs or ECG parameters.
* Subject is electrically sensitive (e.g., prior iontophoresis with adverse outcome related to the current delivered by the device) or who have an implantable electronic device (e.g., pacemaker).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Analysis of variance (ANOVA) will be used to compare AUC0-inf and Cmax values between treatments. AUC0-last, Tmax and t1/2 will be summarized descriptively. | Blood samples (4 mL per sample) for PK analysis will be collected for all treatments by catheter or venipuncture into EDTA collection tubes for the determination of sumatriptan concentrations in plasma for each treatment.
  Blood samples (4 mL per sample) for PK analysis will be collected at the following times for the determination of sumatriptan concentrations in plasma for each treatment:
  Pre-dose (within 15 minutes prior to dosing) and at 0.25, 0.50, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hrs post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Canas, MD, Principal Investigator — Prism Research LLC
Locations (1):
- Prism Research, LLC, Saint Paul, Minnesota, United States